CLINICAL TRIAL: NCT03250104
Title: Antibiotic Stewardship and Infection Control in Patients at High Risk of Developing Infection by Clostridium Difficile, Vancomycin-Resistant Enterococci or Multi-Resistant Gram-Negatives
Acronym: ABSOLUTE
Status: Completed | Type: Observational
Sponsor: University Hospital of Cologne (Other)
Collaborators: Charite University, Berlin, Germany (Other); University Hospital Freiburg (Other); University of Hamburg-Eppendorf (Other); University Hospital Lübeck (Other); University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. med. Jörg Janne Vehreschild, Professor, University Hospital of Cologne
Other Study IDs: TTU HAARBI 8.810
Record Dates: First submitted 2017-06-27; First posted 2017-08-15 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Clostridium Difficile Infection; VRE Infection; Nosocomial Infection; MRGN Bacteria
Keywords: antimicrobial stewardship; infection control; nosocomial infection; clostridium difficile; MRGN bacteria; health-care associated pathogens; VRE
MeSH Terms: conditions — Clostridium Infections; Cross Infection | interventions — Infection Control; Antimicrobial Stewardship

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Infection Control — The infection control bundle will include staff training, hand hygiene programs, disinfection measures, and contact isolation. Physicians will be discouraged to prescribe proton pump inhibitors (PPIs) where not explicitly needed. The intervention bundle will be defined based on current literature. For implementation, the investigator will adapt the bundle to specific local needs, discuss with the responsible department heads and ward staff, perform training and disseminate standards of care.
Other: Antibiotic Stewardship — Antibiotic stewards will develop local standards of procedure based on the provided training and guidelines. They will then train the responsible staff and disseminate guidelines as best suited for the local work environment, e.g. as pocket cards, posters, or electronically. Point-prevalence investigations and "antibiotic visits" will assure adherence to guidelines.

SUMMARY:
Throughout project, the investigators design, evaluate and disseminate infection control and antibiotic stewardship (ABS) measures aimed at reducing the incidence of Clostridium difficile infection (CDI). The measures will focus on known departments with high incidence of CDI, i.e. a) hematology/oncology, b) other departments/wards demonstrating above-average infection rates, which were identified throughout previous studies. The infection control package will include staff training, hand hygiene programs and disinfection measures. Throughout the ABS package, investigators will develop and implement ABS measures specifically designed for patients at the highest risk of developing hospital-acquired infections, i.e. those treated on hematological/oncological wards. Potentially useful ABS actions even in critically ill patients are early reduction of exposure based on microbiological results, timely cessation of anti-infective treatment, thoughtful implementation of screening measures and biomarkers, defined approaches to patients known to be allergic to penicillins, and vigorous enforcement of clinical and microbiological diagnosis of infection focus.

The IC and ABS measures aim at educating and assisting clinical personnel in realizing treatments according to official guidelines. There will not be a direct contact between study personnel and patient. There will be no direct recruitment of patients.

DETAILED DESCRIPTION:
In recent years, a distinct group of healthcare-associated pathogens (HPs) has become highly prevalent among hospital inpatients worldwide. Clostridium difficile, vancomycin-resistant enterococci (VRE), and multi-resistant gram-negative bacteria (MRGN) today are an immediate threat to hospitalized patients in Western countries, given inferior outcomes and prolonged treatment associated with such infections.

There are two key clinical strategies to prevent transmission and reduce the overall incidence of infections by Clostridium difficile and other gut-derived HPs. Infection control (IC) measures act by avoiding in-hospital transmissions using various interventions, including hand hygiene, contact isolation and environmental cleaning/disinfection. Antibiotic stewardship (ABS) on the other hand aims at reducing selective pressure by ascertaining adequacy of treatment duration, dose, and selection of antibiotics.However, there is a scarcity of studies showing effectiveness of these strategies in actually reducing nosocomial infection by HPs. Single room contact isolation has deleterious implications, i.e. increased cost, decreased patient contacts and quality of life, but has not been proven effective for most HPs. Current ABS concepts are usually not aimed at the patients with the highest antibiotic consumption and the highest risk of contracting nosocomial infection by HPs, e.g. patients with neutropenia following chemotherapy.

ABSOLUTE is a comprehensive clinical study programme assessing IC/ABS measures to reduce Clostridium difficile infections (CDI) on high-incidence HP/CDI wards in a stepped-wedge cluster-randomized trial. The study will focus on known departments with high incidence of CDI, i.e. a) hematology/oncology, b) other departments/wards demonstrating above-average infection rates, which will be identified throughout previous study by the German Center for Infection Research (DZIF). This design was chosen as high-risk groups allow optimal resource utilization by expedited observation of target outcomes and because there is a translational gap towards implementing established strategies of infection control and ABS in critically ill patient groups.

Each partner site will identify eight observation wards. To allow measurement of secondary endpoints relevant to the IC/ABS bundle, especially safety, at least three of the sites should include their hematology/oncology department into the analysis. The other wards/departments will be selected based on CDI epidemiology. Incidence of CDI on candidate study wards/departments should exceed the 75 percentile based on R-Net (DZIF study) data collected during the preparation phase. The study coordinators will make the ultimate decision on the participating wards based on discussion with the local team of investigators. Besides the above-mentioned entry criteria, knowledge of current practices and approachability of the ward and the related staff may be regarded during the discussion. In total, each site will perform the analysis on at least ten wards of at least three departments.

Infection control measures for Clostridium difficile are well established and can be easily applied into hospital routine. This work package can therefore start ahead of the ABS bundle with measures aimed at reducing transmission of Clostridium difficile. The infection control bundle will include staff training, hand hygiene programs, disinfection measures, and contact isolation. Physicians will be discouraged to prescribe proton pump inhibitors (PPIs) where not explicitly needed. The bundle will be defined based on current literature. During the preparation phase of the study, investigators and other personnel from each site will receive central training courses in infection control measures targeted at reduction of effective Clostridium difficile transmission. It will be their task to train local staff (ward physicians, nurses) for compliance with the infection control bundle. For implementation, the investigator will adapt the bundle to specific local needs, discuss with the responsible department heads and ward staff, perform training and disseminate standards of care. The following indicators of process quality will be measured be the investigator in collaboration with the local hygiene staff: compliance observations (contact isolation, hand hygiene), education assessment (surveys), and PPI consumption.

Throughout the ABS work package, the investigators will develop and implement an ABS bundle specifically designed for patients at the highest risk of developing hospital-acquired infections, i.e. those treated on hematological/oncological wards. Potentially useful ABS measures even in critically ill patients are early reduction of exposure based on microbiological results, timely cessation of anti-infective treatment, thoughtful implementation of screening measures and biomarkers, defined approaches to patients known to be allergic to penicillins, and vigorous enforcement of clinical and microbiological diagnosis of infection focus. The study hypothesis is, that the consumption of glycopeptides, carbapenems, daptomycin, tigecycline, and linezolid can be significantly reduced without jeopardizing patient outcomes. Reduction of these antibiotics will save last resort antimicrobials for documented breakthrough infections, reduce colonization and blood stream infections (BSI) with VRE and extended-spectrum beta-lactamase-producing gram-negatives (ESBL), and reduce the incidence of CDI.

As a first step, the investigators will guide a consensus process to develop specific ABS guidelines for hematology/oncology wards. They will develop this guideline primarily as German S2k (consensus) guideline, but will also seek publication in an international peer-reviewed journal. For the consensus process, relevant German medical societies and groups will be invited to send delegates. External experts will be invited to participate in the process and comment on the guideline as needed. The consensus process will consist of a kick-off face-to-face meeting with discussion and distribution of work packages, monthly telephone conferences and finally, a consensus meeting. The guidelines will contain advice on specific strategies to avoid excessive or wrong usage of anti-infectives and also on quality indicators of appropriate antibiotic use.

All study sites will receive comprehensive training in the defined ABS criteria as part of a 3-day course program. In addition, sites without established ABS groups or trained ABS experts will receive standard three-week training by the ABS Initiative (www.antibiotic-stewardship.de). Afterwards, implementation of the ABS measures will start. Antibiotic stewards will develop local standards of procedure based on the provided training and guidelines. They will then train the responsible staff and disseminate guidelines as best suited for the local work environment, e.g. as pocket cards, posters, or electronically. Point-prevalence investigations will assure adherence to guidelines.

ELIGIBILITY:
Inclusion Criteria:

- patients admitted to departments with high incidence of CDI, i.e. a) hematology/oncology, b) other departments/wards demonstrating above-average infection rates (identified by previous studies)

Exclusion Criteria:

- patients admitted in opthalmology, paediatrics, psychiatry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted on wards with high incidence of CDI.
Sampling Method: Non-Probability Sample
Enrollment: 80000 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
CDI incidence | Baseline and every 3 months up to 144 weeks
  Significant reduction of the overall CDI incidence on intervention wards following implementation of the combined IC and ABS bundles in pre-post analysis stratified by center.

SECONDARY OUTCOMES:
Effectiveness of IC bundle through incidence of CDI or BSI by VRE and MRGN | Baseline and every 3 months up to 144 weeks
  Effectiveness of the infection control bundle for preventing nosocomial infection by incidence of a) CDI, or BSI by b) VRE, and c) MRGN by pre-post analysis before implementation of the ABS bundle.
PPI usage | Baseline and every 3 months up to 144 weeks
  Reduction in the consumption of PPIs, measured by Defined Daily Dose (DDD) before and after IC bundle implementation
Improvement of process indicators by calculating disinfectant consumption and antibiotic consumption | Baseline and every 3 months up to 144 weeks
  Improvement of process indicators for the IC (disinfectant consumption) and ABS (antibiotic consumption) bundles by pre-post analysis before implementation of the measures
Effectiveness of ABS interventions by continuously measuring RDDs | Baseline and every 3 months up to 144 weeks
  Effectiveness of ABS interventions in reducing consumption of antibiotics discouraged for empirical treatment (3rd generation cephalosporins, glycopeptides, carbapenems, daptomycin, tigecycline, and linezolid), measured by Recommended Daily Dose (RDDs) before and after ABS bundle implementation
Antibiotic consumption | Baseline and every 3 months up to 144 weeks
  Time series analysis using monthly aggregations of antibiotic consumption (RDDs) and incidence of a) CDI, b) VRE, and c) MRGN on participating wards and correlation with IC and ABS intervention activities
Cost-effectiveness by comparing expenditures of implementing IC/ABS measures with reduction in antibiotic consumption | Baseline and after 144 weeks (end of the study)
  Cost-effectiveness of the different bundles by reducing antibiotic consumption, abbreviating average inpatient stays, and reducing the need for intensive care treatment compared to expenditure for IC and ABS bundle implementation

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Janne Vehreschild, MD, Principal Investigator — University Hospital Cologne
Locations (1):
- University Hospital of Cologne, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared after the end of the study

REFERENCES:
- [Background] Gastmeier P, Weitzel-Kage D, Behnke M, Eckmanns T. Surveillance of Clostridium difficile-associated diarrhoea with the German nosocomial infection surveillance system KISS (CDAD-KISS). Int J Antimicrob Agents. 2009 Mar;33 Suppl 1:S19-23. doi: 10.1016/S0924-8579(09)70011-1. PMID 19303563
- [Background] Meyer E, Gastmeier P, Weizel-Kage D, Schwab F. Associations between nosocomial meticillin-resistant Staphylococcus aureus and nosocomial Clostridium difficile-associated diarrhoea in 89 German hospitals. J Hosp Infect. 2012 Nov;82(3):181-6. doi: 10.1016/j.jhin.2012.07.022. Epub 2012 Sep 27. PMID 23021304
- [Background] Vonberg RP, Kuijper EJ, Wilcox MH, Barbut F, Tull P, Gastmeier P; European C difficile-Infection Control Group; European Centre for Disease Prevention and Control (ECDC); van den Broek PJ, Colville A, Coignard B, Daha T, Debast S, Duerden BI, van den Hof S, van der Kooi T, Maarleveld HJ, Nagy E, Notermans DW, O'Driscoll J, Patel B, Stone S, Wiuff C. Infection control measures to limit the spread of Clostridium difficile. Clin Microbiol Infect. 2008 May;14 Suppl 5:2-20. doi: 10.1111/j.1469-0691.2008.01992.x. PMID 18412710
- [Background] Vehreschild MJ, Hamprecht A, Peterson L, Schubert S, Hantschel M, Peter S, Schafhausen P, Rohde H, Lilienfeld-Toal MV, Bekeredjian-Ding I, Libam J, Hellmich M, Vehreschild JJ, Cornely OA, Seifert H. A multicentre cohort study on colonization and infection with ESBL-producing Enterobacteriaceae in high-risk patients with haematological malignancies. J Antimicrob Chemother. 2014 Dec;69(12):3387-92. doi: 10.1093/jac/dku305. Epub 2014 Aug 6. PMID 25103492
- [Background] Vehreschild MJ, Weitershagen D, Biehl LM, Tacke D, Waldschmidt D, Tox U, Wisplinghoff H, Von Bergwelt-Baildon M, Cornely OA, Vehreschild JJ. Clostridium difficile infection in patients with acute myelogenous leukemia and in patients undergoing allogeneic stem cell transplantation: epidemiology and risk factor analysis. Biol Blood Marrow Transplant. 2014 Jun;20(6):823-8. doi: 10.1016/j.bbmt.2014.02.022. Epub 2014 Mar 6. PMID 24607558
- [Background] Borde JP, Litterst S, Ruhnke M, Feik R, Hubner J, deWith K, Kaier K, Kern WV. Implementing an intensified antibiotic stewardship programme targeting cephalosporin and fluoroquinolone use in a 200-bed community hospital in Germany. Infection. 2015 Feb;43(1):45-50. doi: 10.1007/s15010-014-0693-2. Epub 2014 Oct 25. PMID 25344419
- [Background] Borde JP, Kaier K, Steib-Bauert M, Vach W, Geibel-Zehender A, Busch H, Bertz H, Hug M, de With K, Kern WV. Feasibility and impact of an intensified antibiotic stewardship programme targeting cephalosporin and fluoroquinolone use in a tertiary care university medical center. BMC Infect Dis. 2014 Apr 15;14:201. doi: 10.1186/1471-2334-14-201. PMID 24731220
- [Background] Vehreschild JJ, Bohme A, Cornely OA, Kahl C, Karthaus M, Kreuzer KA, Maschmeyer G, Mousset S, Ossendorf V, Penack O, Vehreschild MJGT, Bohlius J. Prophylaxis of infectious complications with colony-stimulating factors in adult cancer patients undergoing chemotherapy-evidence-based guidelines from the Infectious Diseases Working Party AGIHO of the German Society for Haematology and Medical Oncology (DGHO). Ann Oncol. 2014 Sep;25(9):1709-1718. doi: 10.1093/annonc/mdu035. Epub 2014 Mar 14. PMID 24631945
- [Background] Vehreschild JJ, Morgen G, Cornely OA, Hartmann P, Koch S, Kalka-Moll W, Wyen C, Vehreschild MJ, Lehmann C, Gillor D, Seifert H, Kremer G, Fatkenheuer G, Jung N. Evaluation of an infectious disease consultation programme in a German tertiary care hospital. Infection. 2013 Dec;41(6):1121-8. doi: 10.1007/s15010-013-0512-1. Epub 2013 Aug 8. PMID 23925637